CLINICAL TRIAL: NCT03996486
Title: A Multicenter, Non-randomized, Open-label, Multiple Dose Escalation Study to Evaluate the Safety and Tolerability of Subcutaneous BAY1093884 in Males With Severe Hemophilia
Brief Title: Study to Test the Safety of an Investigational Drug Given Repeatedly to Adult Men With Severe Hemophilia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Company decision
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 20414; 2018-004566-34 (EudraCT Number)
Record Dates: First submitted 2019-06-21; First posted 2019-06-24 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Hemophilia
Keywords: Coagulation Factor VIII (FVIII); Coagulation Factor IX (FIX); Anti-tissue factor pathway inhibitor (aTFPI); Human monoclonal immunoglobulin G2 antibody
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hemophilia (Experimental): Dose escalation starting with 200 mg of BAY1093884
  Interventions: Drug: BAY1093884

INTERVENTIONS:
Drug: BAY1093884 — Drug administered via subcutaneous injections once weekly for 6 weeks (= 6 doses)
  Other Names: Human monoclonal immunoglobulin G2 antibody blocking the endogenous tissue factor pathway inhibitor (TFPI)

SUMMARY:
The purpose of this study is to investigate the safety of a test drug to treat hemophilia in adult men.

DETAILED DESCRIPTION:
The primary objective is to assess the safety of multiple doses of BAY1093884.

ELIGIBILITY:
Inclusion Criteria:

* Participants with hemophilia A and FVIII activity <1% or hemophilia B with FIX activity <2%
* Participants must be currently without inhibitors or with low titer inhibitors (inhibitor titer < 5 Bethesda units) who are receiving current on demand treatment with any FVIII or FIX (recombinant or plasma-derived; modified or unmodified)

Exclusion Criteria:

* History or at risk of developing diseases related to venous thromboembolic events (e.g., pulmonary embolism, deep vein thrombosis or thrombophlebitis)
* History of any other clinically relevant coagulation disorder (particularly disseminated intravascular coagulopathy or combined FVIII/Factor V deficiency) or platelet disorder
* History or at risk of developing cardiac, coronary and/or arterial peripheral atherosclerotic disease and/or arterial thromboembolic events, particularly myocardial infarction, cerebrovascular accident, stroke, transient ischemic attack, congestive heart failure, angina pectoris, treatment for angina pectoris or uncontrolled hypertension
* History or at risk for thrombotic microangiopathy

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-28 (Estimated); Primary Completion 2020-05-29 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of drug-related adverse events | Up to 3 months
Frequency of drug-related serious adverse events | Up to 3 months
Frequency of adverse events of special interest | Up to 3 months
  Adverse events of special interest comprise thromboembolic and thrombotic microangiopathy events, and hypersensitivity reactions.

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.